CLINICAL TRIAL: NCT06024993
Title: Dead Space in Mechanical Ventilation With Constant Expiratory Flow
Acronym: DeXFLoW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 003029
Record Dates: First submitted 2023-04-03; First posted 2023-09-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Mechanical Ventilation; Artificial Respiration

STUDY DESIGN:
Intervention Model Description: Crossover volume-controlled ventilation and flow-controlled ventilation
Who Masked: Participant, Outcomes Assessor
Masking Description: During analysis the groups (flow-controlled ventilation and volume-controlled ventilation) will be blinded.
  Participants know that they will be exposed to both modes of ventilation, but are unaware of the randomized sequence (FCV-VCV or VCV-FCV).
  It is impossible to mask the investigators delivering the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FCV-VCV (Experimental): After titration of ventilation in baseline VCV (all arms), participants will first receive 20 min of baseline-matched FCV and subsequently 20 min of baseline-matched VCV.
  Interventions: Device: Flow-controlled ventilation (FCV); Device: Conventional volume-controlled ventilation (VCV)
- VCV-FCV (Experimental): After titration of ventilation in baseline VCV (all arms), participants will first receive 20 min of baseline-matched VCV and subsequently 20 min of baseline-matched FCV.
  Interventions: Device: Flow-controlled ventilation (FCV); Device: Conventional volume-controlled ventilation (VCV)

INTERVENTIONS:
Device: Flow-controlled ventilation (FCV) — 20 minutes of FCV, delivered with the CE-marked Evone ventilator (Ventinova medical, the Netherlands)
Device: Conventional volume-controlled ventilation (VCV) — 20 minutes of conventional VCV, delivered with the CE-marked Aisys CS3 (GE Healthcare, USA) or Flow-i (Getinge, Sweden) ventilators.

SUMMARY:
Conventional continuous mandatory mechanical ventilation relies on the passive recoil of the chest wall for expiration. This results in an exponentially decreasing expiratory flow.

Flow controlled ventilation (FCV), a new ventilation mode with constant, continuous, controlled expiratory flow, has recently become clinically available and is increasingly being adopted for complex mechanical ventilation during surgery.

In both clinical and pre-clinical settings, an improvement in ventilation (CO2 clearance) has been observed during FCV compared to conventional ventilation. Recently, Schranc et al. compared flow-controlled ventilation with pressure-regulated volume control in both double lung ventilation and one-lung ventilation in pigs. They report differences in dead space ventilation that may explain the improved CO2 clearance, although their study was not designed to compare dead space ventilation within the group of double lung ventilation.

Dead space ventilation, or "wasted ventilation", is the ventilation of hypoperfused lung zones, and is clinically relevant, as it is a strong predictor of mortality in patients with the acute respiratory distress syndrome (ARDS) and is correlated with higher airway driving pressures which are thought to be injurious to the lung (lung stress).

This trial aims to study the difference in dead space ventilation between conventional mechanical ventilation in volume-controlled mode and flow controlled-ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults [18-70] yrs
* General anaesthesia for elective surgery
* Arterial line, central venous line and endotracheal tube as part of standard of care
* Expected duration of controlled mechanical ventilation ≥ 60 minutes
* Supine position (0±10°)

Exclusion Criteria:

* One lung ventilation
* Known pregnancy
* Increased intra-abdominal pressure (pneumoperitoneum or obesity (BMI > 30kg/m2))
* COPD GOLD IV or home oxygen dependence
* Cardiac pacemaker, implantable cardioverter-defibrillator (ICD) or thoracic neurostimulator
* Skin lesions (e.g. injury, inflammation) at the level where the Electrical Impedance Tomography (EIT) band is to be applied
* Clinical signs of raised intracranial pressure
* Potential interference with the surgery due to the setup of the study instruments.
* Patient refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Bohr dead space ventilation (VDBr/VT) | During FCV and VCV measurements (20 minutes)
  Quantified by the Bohr approach with volumetric capnography

SECONDARY OUTCOMES:
Change in Enghoff dead space ventilation (VDEng/VT) | During FCV and VCV measurements (20 minutes)
  Quantified by the Enghoff approach with volumetric capnography
Change in physiological dead space volume (Vdfys) | During FCV and VCV measurements (20 minutes)
  Measured with volumetric capnography and Enghoff's approach
Change in airway dead space volume (Vdaw) | During FCV and VCV measurements (20 minutes)
  Measured with volumetric capnography and Fletcher's approach
Change in alveolar dead space volume (Vdalv) | During FCV and VCV measurements (20 minutes)
  As measured with volumetric capnography and Fletcher's approach
Ventilatory efficiency (VE/VCO2) | During FCV and VCV measurements (20 minutes)
  Ratio of minute ventilation to carbon dioxide output
Change in airway driving pressure (∆Paw) | During FCV and VCV measurements (20 minutes)
  Calculated as the difference between the plateau pressure (Pplat) during an inspiratory pause and the dynamic positive end-expiratory pressure (PEEP), as no expiratory hold is possible on the Evone.
Change in transpulmonary shunt fraction (Qs/Qt) | During FCV and VCV measurements (20 minutes)
  calculated with the modified Berggren equation
Change in global lung hyperdistention (hyperdistentionEIT) | During FCV and VCV measurements (20 minutes)
  Calculated from electric impedance tomography
Change in anterio-posterior distribution of ventilation on EIT (AP) | During FCV and VCV measurements (20 minutes)
  % anterior / % posterior
Change in right-left distribution of ventilation on EIT (RL) | During FCV and VCV measurements (20 minutes)
  % right / % left
Change in 4-layered distribution of ventilation on EIT | During FCV and VCV measurements (20 minutes)
Change in centre of ventilation on EIT | During FCV and VCV measurements (20 minutes)
Change in cardiac index (CI) | During FCV and VCV measurements (20 minutes)
  Calculated from the arterial waveform (pulse contour analysis) by the HemoSphere monitor
Change in mean arterial pressure (MAP) | During FCV and VCV measurements (20 minutes)
  Measured on a radial artery line
Change in partial pressure of arterial CO2 (PaCO2) | During FCV and VCV measurements (20 minutes)
  Measured on an arterial blood gas
Change in peak expiratory flow (PEF) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in peak inspiratory flow (PIF) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in mean airway pressure (MPaw) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in tidal volume (TV) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in respiratory rate (RR) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in minute ventilation (MV) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in inspiratory time (Ti) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in expiratory time (Te) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in ratio of inspiratory time to total breath time (Ti / Tt) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in positive end-expiratory pressure (PEEP) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in peak inspiratory pressure (PIP) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in plateau pressure (Pplat) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in static airway compliance (Caw) | During FCV and VCV measurements (20 minutes)
  Calculated as tidal volume / airway driving pressure
Change in end-tidal CO2 (ETCO2) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in global airway resistance (Raw) | During FCV and VCV measurements (20 minutes)
  As measured by the citrex respiratory monitor
Change in global airway time constant (TAUaw) | During FCV and VCV measurements (20 minutes)
  Calculated as global airway resistance x global airway compliance
Change in total energy | During FCV and VCV measurements (20 minutes)
  As calculated from monitoring data
Change in dissipated energy | During FCV and VCV measurements (20 minutes)
  As calculated from monitoring data
Change in P/F ratio | During FCV and VCV measurements (20 minutes)
  Calculated as partial pressure of arterial oxygen divided by inspiratory fraction of oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, M.D., Ph.D., Principal Investigator — Antwerp University Hospital / University of Antwerp
Locations (1):
- Antwerp University Hospital (UZA), Edegem, Antwerp, Belgium